CLINICAL TRIAL: NCT00738491
Title: Effects of Ambient Air Pollution Exposure in Patients With Stable Angina Pectoris During Normal Daily Activities
Status: Terminated | Type: Observational
Why Stopped: Study performed in alternative location (Beijing China)
Sponsor: University of Edinburgh (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Jeremy Langrish, Clinical Lecturer and Specialty Registrar in Cardiology, University of Edinburgh
Other Study IDs: 08/S1101/6
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Angina Pectoris; Coronary Heart Disease
Keywords: Angina pectoris; Exercise capacity; Myocardial ischaemia; Air pollution
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with stable angina pectoris and documented coronary heart disease recruited in Edinburgh
- 2: Patients with stable angina pectoris and documented coronary heart disease recruited in London

SUMMARY:
The purpose of this study is to identify whether exposure to ambient levels of air pollution during normal daily activities has a functional impact on patients with coronary heart disease

DETAILED DESCRIPTION:
Exposure to air pollution has been shown in epidemiological studies to be closely linked to cardiovascular morbidity and mortality. The exact components of air pollution that underlie the cardiovascular effects are not yet known, but combustion-derived particulate matter is suspected to be the major cause. In controlled exposure studies, we have recently demonstrated that exposure to diesel exhaust causes increased myocardial ischaemia with exercise in patients with asymptomatic coronary artery disease. The mechanism behind this effect is not yet understood, but we have shown that diesel exhaust exposure causes an acute impairment of two important and highly relevant aspects of vascular tone: vasomotor tone and endogenous fibrinolysis. In this study we propose to investigate the effects of exposure to ambient levels of air pollution on patients with stable, symptomatic angina pectoris, during their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Documented coronary artery disease
* Symptoms of stable angina pectoris
* Positive BRUCE exercise stress test between 3 and 13 minutes

Exclusion Criteria:

* History of arrhythmia
* Severe 3 vessel coronary disease or left main stem stenosis that has not been revascularised
* Resting conduction abnormality
* Digoxin therapy
* Uncontrolled hypertension
* Renal or hepatic failure
* Unstable symptoms or acute coronary syndrome within 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stable angina pectoris and documented coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Symptoms of angina pectoris - assessed by symptom diary and reliever medication usage | Throughout study period

SECONDARY OUTCOMES:
Myocardial ischaemic burden - assessed using 12-lead continuous Holter ECG monitoring | Throughout study period
Time to 1mm ST segment depression during standard BRUCE exercise stress testing | At the end of the study period
Total exercise capacity - measured using GPS tracking of activity completed | Throughout study period
Exercise capacity - determined by standard BRUCE exercise stress testing | Immediately after study period
Ambulatory blood pressure | Throughout study period
Biochemical evidence of myocardial ischaemia - highly sensitive troponin, ischaemically modified albumin and fatty acid binding protein | Before and after study period

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Langrish, MB BCh, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - University of Edinburgh, Edinburgh, Midlothian
  - Imperial College, London

REFERENCES:
- [Background] McCreanor J, Cullinan P, Nieuwenhuijsen MJ, Stewart-Evans J, Malliarou E, Jarup L, Harrington R, Svartengren M, Han IK, Ohman-Strickland P, Chung KF, Zhang J. Respiratory effects of exposure to diesel traffic in persons with asthma. N Engl J Med. 2007 Dec 6;357(23):2348-58. doi: 10.1056/NEJMoa071535. PMID 18057337
- [Background] Mills NL, Tornqvist H, Gonzalez MC, Vink E, Robinson SD, Soderberg S, Boon NA, Donaldson K, Sandstrom T, Blomberg A, Newby DE. Ischemic and thrombotic effects of dilute diesel-exhaust inhalation in men with coronary heart disease. N Engl J Med. 2007 Sep 13;357(11):1075-82. doi: 10.1056/NEJMoa066314. PMID 17855668
- [Background] Tornqvist H, Mills NL, Gonzalez M, Miller MR, Robinson SD, Megson IL, Macnee W, Donaldson K, Soderberg S, Newby DE, Sandstrom T, Blomberg A. Persistent endothelial dysfunction in humans after diesel exhaust inhalation. Am J Respir Crit Care Med. 2007 Aug 15;176(4):395-400. doi: 10.1164/rccm.200606-872OC. Epub 2007 Apr 19. PMID 17446340
- [Background] Mills NL, Tornqvist H, Robinson SD, Gonzalez M, Darnley K, MacNee W, Boon NA, Donaldson K, Blomberg A, Sandstrom T, Newby DE. Diesel exhaust inhalation causes vascular dysfunction and impaired endogenous fibrinolysis. Circulation. 2005 Dec 20;112(25):3930-6. doi: 10.1161/CIRCULATIONAHA.105.588962. PMID 16365212